CLINICAL TRIAL: NCT04680754
Title: The Effect of Head-Neck Stretching Exercises After Thyroidectomy on Postoperative Pain Level and Wound Healing- Randomised Controlled Trial
Brief Title: The Effect of Head-Neck Stretching Exercises After Thyroidectomy on Postoperative Pain Level and Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acelya Turkmen (Other)
Responsible Party: Sponsor-Investigator, Acelya Turkmen, Research Assistant PhD, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/1763
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain; Postoperative Wound Complication
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study to determine the effect of post-thyroidectomy head-neck stretching exercises on postoperative pain level and wound healing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Routine nursing care (use of analgesics, IV fluid therapy and wound care) was applied to patients in experimental group after thyroidectomy. A brochure was developed in line with the literature on head-neck stretching exercises. Since the patients came to the clinic on surgery day, the exercises were examined by the patient on the first postoperative day. The patient was asked to perform the exercises 3 times a day, in the morning, noon and evening for a month, provided that each movement was 5 times. Then, the "Patient and Observer Scar Rating Scale (POSAS) " was applied.
  The pain level of the patient on postoperative day 1 was evaluated using VAS. For further evaluations, the patient was called by phone at the 1st week and 1st month. Neck pain and discomfort status was evaluated with the "Neck Pain and Disability Scale" (NPAD), and then the scar appearances with the "Patient and Observer Scar Assessment Scale" by requesting neck photographs at the 1st week and 1st month.
  Interventions: Other: head-neck stretching exercises
- Control Arm (No Intervention): Routine nursing care (use of analgesics, IV fluid therapy and wound care) was applied to the control group after thyroidectomy. Follow-up of the patients with the scales applied in the experimental group were also performed to the control group at the same intervals. After thyroidectomy, patients were called by phone in the 1st week and 1st month. "Neck pain and discomfort scale" and "Patient and Observer Scar Rating Scale" were applied again in both phone calls. Photographs of the scar appearance at the 1st week and the 1st month were requested from the patients.

INTERVENTIONS:
Other: head-neck stretching exercises — Neck stretching exercises which include basic movements of the neck are simple and effective exercises. Stretching exercises provide neuromuscular coordination and flexibility in patients by reducing pain and muscle weakness (Nakamura, Kodama, and Mukaino 2014). For this reason, neck stretching exercises should be performed in early postoperative period and a nurse should teach the patient the head-neck stretching exercises and ensure the patient's comfort after thyroidectomy.
  Arms: Experimental Arm

SUMMARY:
Background: Thyroid diseases are one of the most common health problems all over the world. After thyroidectomy, patients often experience discomfort such as neck pain, shoulder stiffness, shoulder movement difficulty, choking or pressing feeling. Head-neck stretching exercises provide neuromuscular coordination and flexibility in patients by reducing pain and muscle weakness.

Methods: This research was carried out as a pre-test / post-test control group experimental design study in 82 patients in the general surgery clinic of a university hospital in Istanbul

DETAILED DESCRIPTION:
Thyroid hormones are responsible for many metabolic activities in human physiology. It increases the basal metabolic rate, affects protein synthesis and helps growth of long bones. However, when thyroid functions change in the human body, the individual can be negatively affected and some individuals may require surgical intervention. Thyroid surgery is a prominent treatment for goiter, hyperthyroidism, thyroid nodules or thyroid carcinoma.

It has been reported that the most important complications after thyroidectomy are laryngeal nerve damage and hypoparathyroidism. Therefore, patients generally suffer from uncomfortable symptoms such as neck pain, shoulder stiffness, difficulty moving shoulders, choking or pressing feeling. In addition, it is indicated that in the early postoperative period, patients experience limitation in neck movement and have a robotic walking style in order to prevent possible neck pain and protect the incision area. It is emphasized that these symptoms persist for a while after the operation and negatively affect the daily life of the patient.

Neck stretching exercises which include basic movements of the neck are simple and effective exercises. Stretching exercises provide neuromuscular coordination and flexibility in patients by reducing pain and muscle weakness. For this reason, neck stretching exercises should be performed in early postoperative period and a nurse should teach the patient the head-neck stretching exercises and ensure the patient's comfort after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Having agreed to participate in the research verbally and in writing after being informed about the research,
* 18 years of age or older,
* Patients who were able to understand the information given, who could read, write and speak in Turkish, who have not any problems preventing verbal communication, and who underwent thyroid surgery were included in the study.

Exclusion Criteria:

- Patients who suffers from cervical problems before surgery were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | Reported pain severity in the first 24 hours after surgery.
  Pain intensity assesment with Visual Assesment Scale (VAS) Score: 0-10; 0- No pain, 10- Worst pain
Change from Postoperative Neck Pain and Disability at 1 month | Postoperative 1 st week and 1 st mounth
  Neck Pain and Disability Scale (NPDS) The scale consists of 15 items. Each item measures the severity of pain, and evaluates the interaction of professional, social and functional aspects of life, and the presence and extent of emotional factors. Each item has a 10 cm visual analog scale. It is divided into 6 sections at equal intervals by vertical bars. Each item is between 0-5 points.
Change from Postoperative Wound Healing at 1 month | Postoperative 1 st day, 1 st week and 1 st mounth
  Patient and Observer Scar Rating Scale (POSAS) The scale consists of 7 items, 6 of them are for evaluating the scar (pain, itching, color, elasticity, thickness and irregularity assessment) and 1 evaluating the general opinion about the scar. Each item has a Likert-type score ranges from 1 to 10. 1 indicates normal skin, 10 indicates worst scar assessment. The lowest score in scale, which is 6, demonstrates normal skin, the highest score 60 demonstrates the worst possible scar. The scale score is calculated over the first 6 items.

CONTACTS AND LOCATIONS:
Overall Officials: Nihat AKSAKAL, Assoc. Prof. Dr, Study Chair — Istanbul University
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT04680754/Prot_SAP_000.pdf